CLINICAL TRIAL: NCT01956422
Title: Continuous Positive Airway Pressure (CPAP) for Preventing Respiratory Failure After Laparoscopic Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Tommaso Fossali, Consultant, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE#382/2013
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Continuous Positive Airway Pressure [E02.041.625.790.259]; Prostatectomy [E04.950.774.860.625]; Laparoscopy [E01.370.388.250.520]; Pneumoperitoneum [C06.844.670]
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Positive Airway Pressure(CPAP) (Experimental): In the first 24 hours after laparoscopic prostatectomy patients undergo 3 CPAP cycles (PEEP 7.5, FIO2 40% delivered with Helmet)lasting 2 hours.
  Interventions: Device: Continuous Positive Airway Pressure(CPAP)
- Venturi Mask FiO2 40% (Active Comparator): In the first 24 hours after laparoscopic prostatectomy patients breathe Oxygen 40% delivered with Venturi Mask
  Interventions: Device: Venturi Mask FiO2 40%

INTERVENTIONS:
Device: Continuous Positive Airway Pressure(CPAP)
  Arms: Continuous Positive Airway Pressure(CPAP)
Device: Venturi Mask FiO2 40%
  Arms: Venturi Mask FiO2 40%

SUMMARY:
Aim of this study is verify if postoperative CPAP after laparoscopic prostatectomy may reduce the impact of postoperative respiratory failure, defined as occurrence of hypoxemia (PaO2<60 mmHg) and/or reduction of Forced Expiratory Volume in 1 second (FEV1) beyond 70% of basal value.

DETAILED DESCRIPTION:
Laparoscopic radical prostatectomy (LRP) is a wide used, well tolerated procedure. However, the general anesthesia, the need for pneumoperitoneum and Trendelenburg position may have detrimental effects on both pulmonary volumes and mechanics, and they may increase the risk of postoperative respiratory failure (PORF). Continuous positive airway pressure (CPAP) improves oxygenation and reduces the rate of re-intubation in the presence of PORF.

The aim of our study is to investigate postoperative respiratory function and the likely benefits of the use of CPAP, compared with Venturi mask in terms of prevention of post-operative hypoxaemia and worsening of lung spirometry.

CPAP is delivered with "CASTAR" Helmet by StarMed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic prostatectomy
* American Society of Anesthesiologists status I-II

Exclusion Criteria:

* Cardiac functional status New York Heart Association (NYHA) >II
* Chronic Obstructive Pulmonary Disease (COPD) Gold Class >2

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative respiratory failure (PaO2<60mmHg, FEV1<70% of baseline) | 24 hours after the end of surgery

SECONDARY OUTCOMES:
Incidence of pneumonia | Partecipants will be followed for the duration of hospital stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Fossali, Consultant, Principal Investigator — ASST Fatebenefratelli Sacco
Locations (1):
- Ospedale Luigi Sacco, Milan, Lombardy, Italy

REFERENCES:
- [Background] Ferreyra GP, Baussano I, Squadrone V, Richiardi L, Marchiaro G, Del Sorbo L, Mascia L, Merletti F, Ranieri VM. Continuous positive airway pressure for treatment of respiratory complications after abdominal surgery: a systematic review and meta-analysis. Ann Surg. 2008 Apr;247(4):617-26. doi: 10.1097/SLA.0b013e3181675829. PMID 18362624
- [Background] Squadrone V, Coha M, Cerutti E, Schellino MM, Biolino P, Occella P, Belloni G, Vilianis G, Fiore G, Cavallo F, Ranieri VM; Piedmont Intensive Care Units Network (PICUN). Continuous positive airway pressure for treatment of postoperative hypoxemia: a randomized controlled trial. JAMA. 2005 Feb 2;293(5):589-95. doi: 10.1001/jama.293.5.589. PMID 15687314